CLINICAL TRIAL: NCT02988895
Title: A Prospective Study of Episcleral Brachytherapy for the Treatment of Neovascular Age-related Macular Degeneration
Brief Title: Episcleral Brachytherapy for the Treatment of Wet AMD
Acronym: NEAMES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Salutaris Medical Devices, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMD-201601
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Macular Degeneration, Choroidal Neovascularization
Keywords: Brachytherapy; Wet AMD
MeSH Terms: conditions — Choroidal Neovascularization | interventions — Strontium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- episcleral brachytherapy (Experimental): single fraction of 24 Gy Strontium90 episcleral brachytherapy
  Interventions: Radiation: episcleral brachytherapy

INTERVENTIONS:
Radiation: episcleral brachytherapy — The study intervention is an outpatient, ambulatory procedure performed under local anesthesia with anesthesia assist.
  Other Names: Strontium 90

SUMMARY:
This is a prospective, multi-site, safety and feasibility study of the SalutarisMD SMD-DA system for retrobulbar minimally invasive episcleral brachytherapy device in patients receiving and not responding to anti-VEGF therapy for nAMD. The trial will be open label and non-randomized. The study intervention is a one-time intervention and requires no alteration to the standard of care during the follow-up period.

DETAILED DESCRIPTION:
Subjects will receive a single brachytherapy treatment and 36 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active CNV or PCV due to nAMD
* Poor or non-responsive to FDA approved intravitreal anti-VEGF therapy for nAMD
* BCVA 20/63 or worse Snellen equivalent in the study eye
* Ability to understand nature/purpose of trial and to provide informed consent
* Ability to undergo diagnostic tests and surgical interventions
* Ability to follow instructions and complete the trial including all scheduled visits and follow-up

Exclusion Criteria:

* Neovascularization other than due to AMD
* Sub-foveal lesion hemorrhage obscuring >50% of lesion
* Targeted neovascular lesion with greatest linear dimension >3750 microns or <1000 microns as determined by angiography
* Presence of subretinal fibrosis, including disciform scar, or retinal pigment epithelial (RPE) atrophy that is extensive or foveal threatening in the study eye
* An existing retinal pigment epithelial (RPE) tear
* Previous treatment (excluding vitamins) for nAMD in the study eye other than anti-VEGF therapy in the last 6 months
* A change in anti-VEGF agent in the previous two administrations
* Anticipate a change to the anti-VEGF agent during the conduct of the study
* Other clinically significant ocular co-morbidity including, but not limited to, glaucoma, optic neuropathy of any cause, maculopathy / retinopathy of any cause other than nAMD, scleritis, enophthalmos, microphthalmia, or other co-morbidities that in the investigator's opinion could require medical or surgical intervention to prevent or treat visual loss or media opacity that might result from that condition (i.e. severe cataracts).
* Previous intraocular surgery in study eye other than for uncomplicated phacoemulsification cataract extraction
* High myopia indicated by a history of refractive error of - 6D or greater (spherical equivalent), demonstrated myopic degeneration, or axial length of >26.5mm.
* Subjects with orbital structural abnormalities, such as small (axial length <21 mm), deep set globes or other globe dystopias that, in the investigator's clinical judgment, would require a change in the angle of insertion or increase the risk of structural damage from retrobulbar anesthesia, sub-Tenon's anesthesia, or retrobulbar device positioning.
* Media opacity sufficient to preclude adequate fundoscopy, OCT, or angiography
* Uncontrolled systemic diseases (e.g. controlled hypertension is acceptable)
* Type I or type II diabetes mellitus
* Any previous therapeutic radiation to the head or neck or other areas that may have resulted in a radiation dose to the retina.
* On anticoagulation or dual anti-platelet therapy with abnormal coagulation panel results.
* Patient unsuitable for IV or local anesthesia
* Any contraindication to anti-VEGF, fluorescein, indocyanine green, topical and local anesthetics, topical antiseptics, or topical antibiotics to be used during the study
* Active ocular or periocular infection or intraocular inflammation
* Fellow eye with a BCVA of 20/63 Snellen Equivalent or worse, with advanced AMD (neovascular or non-exudative AMD with foveal geographic atrophy), or other vision threatening disease that is not eligible for vision restoring treatment (i.e. inoperable cataracts).
* Fellow eye is receiving anti-VEGF therapy
* Have received any investigational treatment for any indication in the previous 30 days
* Any condition which, in the investigators' opinion, would conflict or otherwise prevent the subject from complying with the required procedures, schedule or other study conduct

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Safety of the study intervention | 26 weeks
  Adverse event assessment
Tolerability of the study intervention | During procedure
  Subject pain score during procedure
Feasibility of the study intervention | 1 day
  Investigator ability to place the device and deliver a therapeutic dose

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - University Retina, Oak Forest, Illinois

IPD SHARING:
Plan to Share IPD: No